CLINICAL TRIAL: NCT02646943
Title: Longitudinal Study of Patients With Chronic Chagas Cardiomyopathy in Brazil (SaMi_Trop Project)
Acronym: SaMi-Trop
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Federal University of Minas Gerais (Other); Federal University of São João del-Rei (Unknown)
Responsible Party: Principal Investigator, Ester Cerdeira Sabino, Associate Professor, University of Sao Paulo
Other Study IDs: 2111129; P50AI098461-02 (NIH)
Record Dates: First submitted 2015-12-27; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Chagas Disease
Keywords: Cohort; Biomarkers; Cardiomyopathy
MeSH Terms: conditions — Chagas Disease; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort of patients with chronic chagas cardiomyopathy: We have established a prospective cohort of 1,959 patients with chronic Chagas cardiomyopathy (CCC) to evaluate if a clinical prediction rule based on electrocardiogram (ECG), Brain Natriuretic Peptide (BNP) levels and other biomarkers can be useful in clinical practice.
  The study is being conducted in 21 cities of the northern part of Minas Gerais state in Brazil, and includes a follow up of at least two years. The baseline evaluation included collection of socio-demographic information, social determinants of health, health-related behaviours, comorbidities, medicines in use, history of previous treatment for Chagas Disease (ChD), symptoms, functional class, quality of life, blood sample collection and ECG.

SUMMARY:
BACKGROUND: Chagas Disease (ChD) remains as one of the most neglected diseases in the world, with 8-10 million infected people and only one marginally effective therapeutic. The lack of good biomarkers for active infection or clinical end-points poses a problem for assessing the performance of new drugs or therapeutic interventions. Among the biomarkers, several studies showed that Brain Natriuretic Peptide (NT-ProBNP) is accurate maker of left ventricular systolic and diastolic dysfunction.

OBJECTIVE: Our long term goal is to establish The Sao Paulo-Minas Gerais Tropical Medicine Research Center (SaMi-Trop) as a Center of Excellence for Neglected Infectious Disease Research in Brazil. The Specific Aims are to begin that process by focusing on Trypanosoma cruzi infection with the goal of finding an array of biomarkers that correlate with parasite persistence and Chagas cardiac disease status that can be used to infer risk of disease progression and death as well used as markers of cure (parasite eradication) or clinical efficacy (stabilize or reverse cardiac damage) of novel drugs

METHOD: The investigators established a prospective cohort of 1,959 patients with chronic Chagas cardiomyopathy (CCC). The study is being conducted in 21 cities of the northern part of Minas Gerais state in Brazil, and includes a follow up of at least two years (baseline and 24 months) . The evaluation included collection of socio-demographic information, social determinants of health, health-related behaviours, comorbidities, medicines in use, history of previous treatment for Chagas Disease (ChD), symptoms, functional class, quality of life, blood sample collection and ECG.

DETAILED DESCRIPTION:
RESEARCH STRATEGY

SIGNIFICANCE

The Sao Paulo-Minas Gerais Tropical Medicine Research Center (SaMi-Trop) consists of a network of collaborating scientists in the States of Minas Gerais and São Paulo which has been established for the purpose of developing and conducting research projects on neglected infectious diseases in Brazil, with an initial focus on Chagas Disease biomarker, discovery and validation. The SaMi-Trop represents a major challenge for focused research in neglected diseases, with knowledge that can be applied in primary health care.

Chronic Chagas Cardiomyopathy (CCC) is the most important clinical presentation of Chagas Disease (ChD), eventually affecting approximately 20% to 30% of those in the chronic phase of the disease. CCC comprises a wide range of manifestations, including heart failure, arrhythmias, heart-blocks, sudden death, thromboembolism and stroke [1]. Clinical presentation typically varies widely according to the degree of myocardial damage and most patients present a mild form of heart disease, frequently characterized only by the presence of asymptomatic abnormalities on the ECG or in other complimentary exams [2]. Nonetheless, when heart failure and/or severe arrhythmias manifest, the prognosis is ominous, with high and premature mortality rates, typically in adult male patients,1 but also in the elderly [3]. Indeed, when compared to patients with idiopathic cardiomyopathy, patients with CCC have poorer survival, irrespective of other clinical and echocardiographic parameters [4].

Thus, the clinical course of Chagas heart disease is variable and identifying patients who are at risk of progressive CCC and dying remains a challenge. Several longitudinal studies performed in patients in the chronic phase of ChD demonstrated that many individual characteristics predict an unfavorable prognosis. This subject was systematically reviewed a few years ago and concluded that most studies were described in insufficient detail and/or lacked minimal standards in reporting results. Results have been somewhat inconsistent in different studies, and the best combination of clinical and laboratory variables predictive of mortality has not yet been established [5].

A potentially helpful score to predict death was developed to permit the stratification of risk in Chagas heart disease [6]. Six independent prognostic factors were identified, and each was assigned a number of points: New York Heart Association class III or IV (5 points), evidence of cardiomegaly on radiography (5 points), left ventricular systolic dysfunction on echocardiography (3 points), non-sustained ventricular tachycardia on 24-hour Holter monitoring or stress testing (3 points), low QRS voltage on electrocardiography (2 points), and male sex (2 points) [6. Patients were classified in three risk groups according to the final score: low risk (0 to 6 points), intermediate risk (7 to 11 points), and high risk (12 to 20 points). In the original study, the 5-year mortality rates for these three groups were 2 percent, 18 percent, and 63 percent, respectively.6 Although the score was successfully validated in independent cohorts, [6,7] some important issues may arise. The derivation of the score is complex and it is not easy to calculate during the medical consultation. To be calculated, the patient must be submitted to several exams and procedures, including clinical examination, ECG, Chest x-ray, echocardiogram and Holter monitoring or stress testing. Most of these tests are not available in the rural areas, where most of ChD patients live.

A simple score, based on widely available and low-cost tests, which could stratify the risk of death without complex calculations, might be useful in the primary care setting, where echocardiograms and Holter monitoring are not widely available. Easily obtained variables, such as clinical features, BNP levels and ECG measurements, are good candidates as biomarkers for developing a new simple predictive rule. Moreover, new biomarkers in blood, related mainly to inflammation and the immune response, such as TNF-alpha, adhesion molecules and other cytokines, may be determined to be potent prognostic factors and may be useful in the future for further improvement in risk stratification in CCC.

METHOD

Design

Non-concurrent prospective open cohort study, with minimal follow-up of two years (baseline and 24 months).

Outcome

Primary: death Secondary: hospitalization due to cardiac conditions; new ECG abnormalities

Study Population

Participants will be selected from patients evaluated by the Tele Minas Saude (TMS), the state Tele Health System. Since the TeleHealth System is currently acting in support of the Primary Care system, these patients are under the care of primary care physicians of the Health Family Strategy, a public primary care program that has a high coverage in the state of Minas Gerais.

The inclusion criteria are to be a client of the TMS TeleHealth System, be >18 years old, have a positive history for T cruzi infection or Chagas disease, have an abnormal ECG and to consent to participating in the research program.

The exclusion criteria include pregnancy or breast feeding, and any severe condition with ominous prognosis that indicates a life expectancy of less than two years.

Sample size for patient accrual

Considering the minimal number of events per variable acceptable in a proportional hazards regression analysis of 10 events per variable,8 and maximal number of studied variables of ten, the number of events would be 100 in the whole study. Since the prediction model has to be developed and validated and the whole sample will be divided in two, the number of events should be 200. For a 2-year follow-up period and annual mortality rate of 5% in CCC (10% in 2 years), the calculated sample size is 2,000 subjects.

Since the TMS Telehealth system performs 25,000 ECGs each month (300,000 a year), that ECG abnormalities typical of CCC are observed in 5% of these exams (1,250), and projecting that 10% of these patients would be recruited and agree to participate in this research program, the calculated sample size of 2,000 patients will be recruited in a 16 months' accrual period.

Follow-up

Follow-up will be conducted on a yearly basis, with standardized interviews and new ECG exams performed after two years of baseline. Vital status and hospitalization will also be ascertained by linkage of the study database with mortality and hospitalization databases of the Ministry of Health.

Recruitment, initial evaluation and measurements

Patients will be recruited from among those that regularly attend the public primary care service of State of Minas Gerais in places served by TMS Telehealth System. This system provides teleconsultation and Electrocardiogram services (TeleECG), including interpretation of all ECGs by a cardiologist in the University Hospital. A standardized simple form is completed before the transmission of the ECG data to the University hospital and the question "Do you know if you have Chagas disease?" will be added to this questionnaire. Those who answer yes to this question and have abnormal ECG will be selected. A second visit of the selected patients will be scheduled for performing a short questionnaire (including the evaluation of the functional class) and for collecting blood samples. Blood samples will be sent to a central laboratory for T. cruzi serology and BNP measurements, which will be done by standard techniques. Other blood samples, including plasma for protein and antibody studies and stabilized whole blood lysates for T cruzi PCR (Polymerase Chain Reaction), DNA, will be stored at -80o C to enable batched testing for other biomarkers.

Electrocardiogram services (TeleECG)

The ECG performed in the town of origin of the patients will be sent to be assessed by the TMS Telehealth System specialists. The Telecardiology activities were developed using a digital electrocardiograph installed in the towns, at the Basic Health Units of the public healthcare system. The examination was always carried out after being requested by a physician. The ECG will be sent using communication software developed by the TMS Telehealth System and will be analyzed by a on-duty cardiologist. The report will be sent to the Primary Care facility and the ECG tracings will be transferred to ECG reading center. In this ECG Reading Center, a software developed by Prof. Peter Mac Farlane, from Glasgow University, will analyzes and codify the ECG (by the Minnesota Code) and compare to the previous ECG, according to a validated algorithm [9]. All abnormal codes will be reviewed by an experienced cardiologist.

Data analysis

The standardized mortality ratio (SMR) analysis and a survival analysis will be conducted. The outcome death is death. Also, a survival analysis considering the secondary outcomes - hospitalization due to cardiac conditions and new ECG abnormalities - will be run. The development and validation of the prognostic model will follow current recommendations, including the division of the sample in derivation and validation sample, and the use of modern methods to evaluate the performance of the model [10,11]. Additionally, descriptive spatial analysis using geographic distribution for the SMR and a Bayesian spatial model for small area data will be run.

Innovation

Beyond the relevance of the main goal of this study, it has many unique and innovative aspects, related to the use of knowledge and infra-structure developed for other projects conducted by our research group:

1. The possibility of testing new biomarkers detected in other branches of this study or in the NIH-sponsored REDS-II/III Chagas disease study.
2. The use of the infrastructure and the logistics of the TMS program, a state-wide TeleHealth System coordinated by the University Hospital in the Brazilian state of Minas Gerais
3. The use of the methodology of linkage between our databases and administrative and mortality databases from the Health Ministry to complement the follow-up of the selected patients
4. A standardized codification system of the ECGs, using the facilities of the ECG Reading Center of the long-term longitudinal study on the health of 15,000 adult public servants from Brazilian Universities (ELSA-Brazil).

New biomarkers ChD has a complex physiopathology and many immunological, inflammatory, autonomic and micro-vascular processes have a role in the development or the progression of the disease [12]. The investigators have described increased levels of macrophage inflammatory protein (MIP-1alpha) and Tumor necrosis factor-alpha (TNF-alpha) in ChD patients, [13-15] and that those patients with more severe forms have more elevated levels [13]. Recently, in the ChD study (REDS-II), were studied 600 ChD patients and 500 controls searching for biomarkers related to the disease and CCC. In a preliminary analysis, several biomarkers including high sensitivity troponin, myoglobin, soluble vascular cell adhesion molecule 1 (sVCAM-1), soluble intracellular cell adhesion molecule (sICAM) and myeloperoxidase showed abnormal patterns in T cruzi seropositive and parasitemic donors and CCC patients. These and other biomarkers, including those identified in the transcriptome analysis are candidates to be studied in the whole cohort of 2,000 CCC patients in TMS program or, alternatively, using nested case-control design.

Tele Minas Saude (TMS) Program, a state-wide public TeleHealth System

The TMS program is a partnership between the Minas Gerais State Health Department and the State Research Agency (FAPEMIG) with six public universities of Minas Gerais: Universidade Federal de Minas Gerais (UFMG), Universidade Federal do Triângulo Mineiro (UFTM), Universidade Estadual de Montes Claros (UNIMONTES), Universidade Federal de Juiz de Fora (UFJF), Universidade Federal de São João del-Rei (UFSJ) and Universidade Federal de Uberlândia (UFU), forming the Teleassistance Network of Minas Gerais. Created from a telehealth pilot project in cardiology (2006), later expanded to other specialties and villages and transformed into permanent telehealth service, subsidized by the state government in 2009 [16-18].

The objective is to support infrastructure projects of state public health, initially deployed to support the Primary Health Care and Family Health Teams [16]. At that stage, had as main objective to assist professionals in their daily work to improve access to specialized services, reducing and qualifying referrals of patients to secondary and tertiary care. The main activities offered are a) duty of teleconsultation offline in various medical specialties, nursing, dentistry, physiotherapy, psychology, pharmacy and nutrition, b) duty in telecardiology to analyze electrocardiograms (ECGs) and provide teleconsultations online for critical clinical cases c) technical support online and offline, d) permanent education through workshops and training and e) continuous monitoring of system operation in the municipalities.

So far, the program was implemented in 608 municipalities in the state corresponding to 732 telehealth sites. The primary care units in the villages were equipped with computers, electrocardiograph, digital printer and digital camera. Universities were equipped with workstations and videoconferencing equipment. Since 2006, over 20,000 teleconsultations were conducted and 600,000 ECGs analyzed by experts. These telehealth activities prevented the displacement of patients in 78% of the cases [16].

Linkage of databases The Brazilian Health System is characterized by coexistence of a universal public health system (70-80% of coverage) and a supplementary private network. Mortality data from all Brazilians and from hospitalizations in the public health system are stored in large databases owned and managed by the Health Ministry. Investigators developed a methodology for searching these databases for specific subjects using probabilistic linkage methods. The probabilistic strategy we developed has high accuracy, with a sensitivity of 90.6% and specificity 100% [19]. This method will be used in a complimentary way to direct follow-up.

ECG Reading Center ECG interpretation is subjected to substantial intra- and inter-observer variability. To overcome this problem, a standardized ECG code was developed 50 years ago 20 and has been widely used in epidemiological studies. The visual classification of the ECG using the Minnesota code, nonetheless, is time consuming. The investigators created a ECG Reading Center for the Elsa study, a 10-year longitudinal cohort study of 15,000 public employees of Brazilian Universities. For this ECG Reading Center, was installed a software developed by Prof. Peter MacFarlane, from Glasgow University, that analyzes, codifies and compares the ECG with previous tracings, according to a validated algorithm [9]. This system will be used in the present project.

Preliminary Studies

Diagnostic and prognostic value of BNP In 2002, investigators described, in a study published by The Lancet, that blood levels of BNP are inversely correlated to the systolic left ventricular (LV) ejection fraction, the most used index of LV function in ChD [21]. In patients with abnormal ECG and/or chest X-Ray, BNP elevation had a positive predictive value of 80% and a negative predictive value of 97% for the detection of patients with depressed left ventricular ejection fraction [21]. This results were confirmed in the following years by several other studies by our research group [22-26]. A diagnostic strategy including ECG and BNP performed better than the classical approach with ECG and chest X-Ray [24]. Moreover, BNP was also a marker of ventricular arrhythmia [26] and diastolic dysfunction [22,27].

More recently, was described that BNP levels were strong predictors of the risk of death [28] and in a cohort of 1,398 indwelling elderly from the city of Bambuí, in the state of Minas Gerais, Brazil [28]. The hazard ratio for death was 1.27 for each unit of log-transformed BNP level (95% confidence interval (CI: 1.11, 1.45) among infected persons, independent of potentially confounding factors. Infected persons with baseline BNP levels in the top quartile had a risk of death twice that of persons in the bottom quartile (hazard ratio = 2.07, 95% CI: 1.29, 3.32). In the same population, was found that BNP alone or in association with atrial fibrillation had prognostic value for stroke mortality in T. cruzi chronically infected older adults [29].

Electrocardiographic measures and prognostic models The ECG is the single most important exam in CCC. Numerous epidemiological studies have shown that patients with a normal ECG have an excellent medium-term survival [30,31]. The greater the number and severity of ECG alterations registered in a same tracing, the more advanced the myocardial damage possibly is, and the worse the prognosis should be [12]. We have shown that the QRS duration is moderately correlated with the LV ejection fraction [32] and that, during the follow-up of these patients, the increase in the duration of the QRS complex and the appearance of new electrocardiographic alterations may help in identifying patients with a significant decrease (of 5% or more) in left ventricle ejection fraction [33].

Based in the well-known prognostic value of LV ejection fraction and the presence of ventricular tachycardia, [5] was proposed an alternative approach to the well established Rassi's score, [34,35] considering only three risk factors: left ventricular ejection fraction < 50%, ventricular tachycardia at either stress testing or Holter monitoring, and QRS > 133 ms at ECG (or filtered QRS > 150 ms at signal-averaged ECG).34,35 Low risk group has zero or one risk factor (5-year mortality: 1%), intermediate risk, two factors (20% mortality), and high risk, all three factors (50% mortality). This simplified prognostic score had an excellent performance in predicting death in a study with 74 months of follow up (c statistic 0.92) and it may be an attractive alternative to the established six-factor score.

More recently, the investigators showed that T-wave amplitude variability (TWV), a sophisticated ECG-derived measure of repolarization variability, is independently related to the risk of death in ChD [36]. They have also studied the prognostic value of several new echocardiographic measures [37-39] which could be of physiopathological and clinical relevance, but are not possible to be used for ambulatory patients in the rural area.

Kaplan-Meier curves demonstrating mortality in Chagas disease patients Classified according to the presence prolonged of QRS > 133 ms at ECG; Classified according to a risk score in which each of the following factors is worth one point: ventricular tachycardia at either stress testing or Holter monitoring, left ventricular ejection fraction < 0.50, QRS > 133 ms at ECG. Low risk group has zero or one risk factors, intermediate risk, two factors, and high risk, all three factors.

Summarizing, although we and others investigators have extensively studied prognostic markers in Chagas disease and CCC, there is no definite simple, low-cost prognostic model available to be used in the primary care setting. Standard ECG and BNP levels are good candidates to be selected in this simplified predictive model.

ELIGIBILITY:
Eligibility Criteria: to be a client of the TMS TeleHealth System, have a positive history for T cruzi infection or Chagas disease, have an abnormal ECG and to consent to participating in the research program.

Exclusion Criteria: The exclusion criteria include pregnancy or breast feeding, and any severe condition with ominous prognosis that indicates a life expectancy of less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected based on the ECG results performed in 2011-12 by the Telehealth Network. Since the TeleHealth System is currently acting in support of the Primary Care system, these patients are under the care of primary care physicians of the Health Family Strategy, a public primary care program that has a high coverage in the state of Minas Gerais.
Sampling Method: Non-Probability Sample
Enrollment: 1959 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Death | 24 months

SECONDARY OUTCOMES:
Changes in the ECG pattern | baseline and 24 months
Hospitalization due to cardiovascular | baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ester C Sabino, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: Yes
The Dataset will be open access for two years at the end of the data collection process (August, 2018). In the meantime, applications to use the data should be made by contacting the researchers of the SaMi-Trop cohort and filling up the application form. The questionnaires and interviewer guides of the baseline will also be available in electronic formats at http://www.ufsj.edu.br/tecnologiasemsaude_pesquisa/projetos.php

REFERENCES:
- [Background] Harrell FE, Jr. Regression modeling strategies with applications to linear models, logistic regression, and survival analysis. New York: Springer, 2001.
- [Background] Steyerberg EW. Clinical Prediction Models. A Practical Approach to Development,Validation, and Updating. New York: Springer, 2009.
- [Background] Rassi A Jr, Rassi A. The art of risk stratification in Chagas' disease. J Cardiovasc Electrophysiol. 2008 Jun;19(6):E40; author reply E41. doi: 10.1111/j.1540-8167.2008.01172.x. Epub 2008 Apr 21. No abstract available. PMID 18462337
- [Background] Nunes MC, Reis RC, Colosimo EA, Ribeiro AL, Barbosa FB, da Silva JL, Botoni FA, Barbosa MM, Rocha MO. Risk estimation approach in Chagas disease is still needed. Int J Cardiol. 2011 Mar 3;147(2):294-6. doi: 10.1016/j.ijcard.2010.12.044. Epub 2010 Dec 30. No abstract available. PMID 21194765
- [Result] Rocha MO, Ribeiro AL, Teixeira MM. Clinical management of chronic Chagas cardiomyopathy. Front Biosci. 2003 Jan 1;8:e44-54. doi: 10.2741/926. PMID 12456332
- [Result] Rocha MO, Teixeira MM, Ribeiro AL. An update on the management of Chagas cardiomyopathy. Expert Rev Anti Infect Ther. 2007 Aug;5(4):727-43. doi: 10.1586/14787210.5.4.727. PMID 17678433
- [Result] Lima-Costa MF, Peixoto SV, Ribeiro ALP. Chagas disease and mortality in old age as an emerging issue: 10 year follow-up of the Bambui population-based cohort study (Brazil). Int J Cardiol. 2010 Nov 19;145(2):362-363. doi: 10.1016/j.ijcard.2010.02.036. PMID 20399519
- [Result] Pereira Nunes Mdo C, Barbosa MM, Ribeiro AL, Amorim Fenelon LM, Rocha MO. Predictors of mortality in patients with dilated cardiomyopathy: relevance of chagas disease as an etiological factor. Rev Esp Cardiol. 2010 Jul;63(7):788-97. doi: 10.1016/s1885-5857(10)70163-8. English, Spanish. PMID 20609312
- [Result] Rassi A Jr, Rassi A, Rassi SG. Predictors of mortality in chronic Chagas disease: a systematic review of observational studies. Circulation. 2007 Mar 6;115(9):1101-8. doi: 10.1161/CIRCULATIONAHA.106.627265. PMID 17339568
- [Result] Rassi A Jr, Rassi A, Little WC, Xavier SS, Rassi SG, Rassi AG, Rassi GG, Hasslocher-Moreno A, Sousa AS, Scanavacca MI. Development and validation of a risk score for predicting death in Chagas' heart disease. N Engl J Med. 2006 Aug 24;355(8):799-808. doi: 10.1056/NEJMoa053241. PMID 16928995
- [Result] Rocha MO, Ribeiro AL. A risk score for predicting death in Chagas' heart disease. N Engl J Med. 2006 Dec 7;355(23):2488-9; author reply 2490-1. doi: 10.1056/NEJMc062580. No abstract available. PMID 17151373
- [Result] Peduzzi P, Concato J, Feinstein AR, Holford TR. Importance of events per independent variable in proportional hazards regression analysis. II. Accuracy and precision of regression estimates. J Clin Epidemiol. 1995 Dec;48(12):1503-10. doi: 10.1016/0895-4356(95)00048-8. PMID 8543964
- [Result] Macfarlane PW, Latif S. Automated serial ECG comparison based on the Minnesota code. J Electrocardiol. 1996;29 Suppl:29-34. doi: 10.1016/s0022-0736(96)80016-1. PMID 9238374
- [Result] Biolo A, Ribeiro AL, Clausell N. Chagas cardiomyopathy--where do we stand after a hundred years? Prog Cardiovasc Dis. 2010 Jan-Feb;52(4):300-16. doi: 10.1016/j.pcad.2009.11.008. PMID 20109600
- [Result] Talvani A, Rocha MO, Barcelos LS, Gomes YM, Ribeiro AL, Teixeira MM. Elevated concentrations of CCL2 and tumor necrosis factor-alpha in chagasic cardiomyopathy. Clin Infect Dis. 2004 Apr 1;38(7):943-50. doi: 10.1086/381892. Epub 2004 Mar 10. PMID 15034825
- [Result] Ferreira RC, Ianni BM, Abel LC, Buck P, Mady C, Kalil J, Cunha-Neto E. Increased plasma levels of tumor necrosis factor-alpha in asymptomatic/"indeterminate" and Chagas disease cardiomyopathy patients. Mem Inst Oswaldo Cruz. 2003 Apr;98(3):407-11. doi: 10.1590/s0074-02762003000300021. Epub 2003 Jul 18. PMID 12886425
- [Result] Lula JF, Rocha MO, Nunes Mdo C, Ribeiro AL, Teixeira MM, Bahia MT, Talvani A. Plasma concentrations of tumour necrosis factor-alpha, tumour necrosis factor-related apoptosis-inducing ligand, and FasLigand/CD95L in patients with Chagas cardiomyopathy correlate with left ventricular dysfunction. Eur J Heart Fail. 2009 Sep;11(9):825-31. doi: 10.1093/eurjhf/hfp105. Epub 2009 Aug 4. PMID 19654138
- [Result] Ribeiro AL, Alkmim MB, Cardoso CS, Carvalho GG, Caiaffa WT, Andrade MV, Cunha DF, Antunes AP, Resende AG, Resende ES. Implementation of a telecardiology system in the state of Minas Gerais: the Minas Telecardio Project. Arq Bras Cardiol. 2010 Jul;95(1):70-8. doi: 10.1590/s0066-782x2010005000060. Epub 2010 Jun 11. PMID 20563526
- [Result] Cardoso CS, Bandeira M, Ribeiro AL, Oliveira GL, Caiaffa WT. [Satisfaction scales with health care to cardiovascular diseases: CARDIOSATIS--patient and team]. Cien Saude Colet. 2011;16 Suppl 1:1401-7. doi: 10.1590/s1413-81232011000700075. Portuguese. PMID 21503491
- [Result] Cardoso CS, Ribeiro AL, Castro RL, Cesar CC, Caiaffa WT. Implementation of a cardiology care program in remote areas in Brazil: influence of governability. Rural Remote Health. 2010 Jul-Sep;10(3):1472. Epub 2010 Sep 8. PMID 20839899
- [Result] Migowski A, Chaves RB, Coeli CM, Ribeiro AL, Tura BR, Kuschnir MC, Azevedo VM, Floriano DB, Magalhaes CA, Pinheiro MC, Xavier RM. Accuracy of probabilistic record linkage in the assessment of high-complexity cardiology procedures. Rev Saude Publica. 2011 Apr;45(2):269-75. doi: 10.1590/s0034-89102011005000012. Epub 2011 Feb 25. PMID 21344122
- [Result] BLACKBURN H, KEYS A, SIMONSON E, RAUTAHARJU P, PUNSAR S. The electrocardiogram in population studies. A classification system. Circulation. 1960 Jun;21:1160-75. doi: 10.1161/01.cir.21.6.1160. No abstract available. PMID 13849070
- [Result] Ribeiro AL, dos Reis AM, Barros MV, de Sousa MR, Rocha AL, Perez AA, Pereira JB, Machado FS, Rocha MO. Brain natriuretic peptide and left ventricular dysfunction in Chagas' disease. Lancet. 2002 Aug 10;360(9331):461-2. doi: 10.1016/S0140-6736(02)09638-1. PMID 12241721
- [Result] Barbosa MM, Nunes Mdo C, Ribeiro AL, Barral MM, Rocha MO. N-terminal proBNP levels in patients with Chagas disease: a marker of systolic and diastolic dysfunction of the left ventricle. Eur J Echocardiogr. 2007 Jun;8(3):204-12. doi: 10.1016/j.euje.2006.03.011. Epub 2006 May 2. PMID 16651029
- [Result] Ribeiro AL, Reis AM, Teixeira MM, Rocha MO. Brain natriuretic peptide in Chagas' disease: further insights. Lancet. 2003 Jul 26;362(9380):333. doi: 10.1016/S0140-6736(03)13990-6. No abstract available. PMID 12892979
- [Result] Ribeiro AL, Teixeira MM, Reis AM, Talvani A, Perez AA, Barros MV, Rocha MO. Brain natriuretic peptide based strategy to detect left ventricular dysfunction in Chagas disease: a comparison with the conventional approach. Int J Cardiol. 2006 Apr 28;109(1):34-40. doi: 10.1016/j.ijcard.2005.05.048. Epub 2005 Jul 14. PMID 16023747
- [Result] Talvani A, Rocha MO, Cogan J, Maewal P, de Lemos J, Ribeiro AL, Teixeira MM. Brain natriuretic peptide and left ventricular dysfunction in chagasic cardiomyopathy. Mem Inst Oswaldo Cruz. 2004 Oct;99(6):645-9. doi: 10.1590/s0074-02762004000600020. Epub 2004 Nov 18. PMID 15558179
- [Result] Talvani A, Rocha MO, Cogan J, Maewal P, de Lemos J, Ribeiro AL, Teixeira MM. Brain natriuretic peptide measurement in Chagas heart disease: marker of ventricular dysfunction and arrhythmia. Int J Cardiol. 2005 Apr 28;100(3):503-4. doi: 10.1016/j.ijcard.2004.06.007. No abstract available. PMID 15837098
- [Result] Oliveira BM, Botoni FA, Ribeiro AL, Pinto AS, Reis AM, Nunes Mdo C, Rocha MO. Correlation between BNP levels and Doppler echocardiographic parameters of left ventricle filling pressure in patients with Chagasic cardiomyopathy. Echocardiography. 2009 May;26(5):521-7. doi: 10.1111/j.1540-8175.2008.00842.x. PMID 19452608
- [Result] Lima-Costa MF, Cesar CC, Peixoto SV, Ribeiro AL. Plasma B-type natriuretic peptide as a predictor of mortality in community-dwelling older adults with Chagas disease: 10-year follow-up of the Bambui Cohort Study of Aging. Am J Epidemiol. 2010 Jul 15;172(2):190-6. doi: 10.1093/aje/kwq106. Epub 2010 Jun 25. PMID 20581155
- [Result] Lima-Costa MF, Matos DL, Ribeiro AL. Chagas disease predicts 10-year stroke mortality in community-dwelling elderly: the Bambui cohort study of aging. Stroke. 2010 Nov;41(11):2477-82. doi: 10.1161/STROKEAHA.110.588061. Epub 2010 Sep 23. PMID 20864663
- [Result] Ribeiro AL, Rocha MO. [Indeterminate form of Chagas disease: considerations about diagnosis and prognosis]. Rev Soc Bras Med Trop. 1998 May-Jun;31(3):301-14. doi: 10.1590/s0037-86821998000300008. Portuguese. PMID 9612022
- [Result] Maguire JH, Hoff R, Sherlock I, Guimaraes AC, Sleigh AC, Ramos NB, Mott KE, Weller TH. Cardiac morbidity and mortality due to Chagas' disease: prospective electrocardiographic study of a Brazilian community. Circulation. 1987 Jun;75(6):1140-5. doi: 10.1161/01.cir.75.6.1140. PMID 3552307
- [Result] Ribeiro AL, Rocha MO, Barros MV, Rodrigues AR, Machado FS. A narrow QRS does not predict a normal left ventricular function in Chagas' disease. Pacing Clin Electrophysiol. 2000 Nov;23(11 Pt 2):2014-7. doi: 10.1111/j.1540-8159.2000.tb07076.x. PMID 11139981
- [Result] Nascimento BR, Araujo CG, Rocha MO, Domingues JD, Rodrigues AB, Barros MV, Ribeiro AL. The prognostic significance of electrocardiographic changes in Chagas disease. J Electrocardiol. 2012 Jan-Feb;45(1):43-8. doi: 10.1016/j.jelectrocard.2011.04.011. Epub 2011 Jun 24. PMID 21704321
- [Result] Ribeiro AL, Cavalvanti PS, Lombardi F, Nunes Mdo C, Barros MV, Rocha MO. Prognostic value of signal-averaged electrocardiogram in Chagas disease. J Cardiovasc Electrophysiol. 2008 May;19(5):502-9. doi: 10.1111/j.1540-8167.2007.01088.x. Epub 2008 Feb 4. PMID 18266670
- [Result] Ribeiro AL, Rocha MO, Terranova P, Cesarano M, Nunes MD, Lombardi F. T-wave amplitude variability and the risk of death in Chagas disease. J Cardiovasc Electrophysiol. 2011 Jul;22(7):799-805. doi: 10.1111/j.1540-8167.2010.02000.x. Epub 2011 Jan 14. PMID 21235679
- [Result] Nunes Mdo C, Rocha MO, Ribeiro AL, Colosimo EA, Rezende RA, Carmo GA, Barbosa MM. Right ventricular dysfunction is an independent predictor of survival in patients with dilated chronic Chagas' cardiomyopathy. Int J Cardiol. 2008 Jul 21;127(3):372-9. doi: 10.1016/j.ijcard.2007.06.012. Epub 2007 Aug 8. PMID 17689706
- [Result] Nunes MC, Barbosa MM, Ribeiro AL, Colosimo EA, Rocha MO. Left atrial volume provides independent prognostic value in patients with Chagas cardiomyopathy. J Am Soc Echocardiogr. 2009 Jan;22(1):82-8. doi: 10.1016/j.echo.2008.11.015. PMID 19131007
- [Derived] Ferreira AM, Santos LI, Sabino EC, Ribeiro ALP, Oliveira-da Silva LC, Damasceno RF, D'Angelo MFSV, Nunes MDCP, Haikal DSA. Two-year death prediction models among patients with Chagas Disease using machine learning-based methods. PLoS Negl Trop Dis. 2022 Apr 14;16(4):e0010356. doi: 10.1371/journal.pntd.0010356. eCollection 2022 Apr. PMID 35421085
- [Derived] Quintino ND, Sabino EC, da Silva JLP, Ribeiro ALP, Ferreira AM, Davi GL, Oliveira CDL, Cardoso CS. Factors associated with quality of life in patients with Chagas disease: SaMi-Trop project. PLoS Negl Trop Dis. 2020 May 27;14(5):e0008144. doi: 10.1371/journal.pntd.0008144. eCollection 2020 May. PMID 32459812
- [Derived] Cardoso CS, Ribeiro ALP, Oliveira CDL, Oliveira LC, Ferreira AM, Bierrenbach AL, Silva JLP, Colosimo EA, Ferreira JE, Lee TH, Busch MP, Reingold AL, Sabino EC. Beneficial effects of benznidazole in Chagas disease: NIH SaMi-Trop cohort study. PLoS Negl Trop Dis. 2018 Nov 1;12(11):e0006814. doi: 10.1371/journal.pntd.0006814. eCollection 2018 Nov. PMID 30383777
- [Derived] Cardoso CS, Sabino EC, Oliveira CD, de Oliveira LC, Ferreira AM, Cunha-Neto E, Bierrenbach AL, Ferreira JE, Haikal DS, Reingold AL, Ribeiro AL. Longitudinal study of patients with chronic Chagas cardiomyopathy in Brazil (SaMi-Trop project): a cohort profile. BMJ Open. 2016 May 4;6(5):e011181. doi: 10.1136/bmjopen-2016-011181. PMID 27147390